CLINICAL TRIAL: NCT04868409
Title: A Single Blinded Multicenter Randomized Study Comparing Intubating Conditions During Rapid Sequence Induction With Either Suxamethonium 1.0 mg/kg or Rocuronium 1.0 mg/kg in Elderly Patients (≥ 80 Years Old)
Brief Title: Intubating Conditions During Rapid Sequence Induction in Elderly With Either Suxamethonium 1.0 mg/kg or Rocuronium 1.0 mg/kg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-20074958
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Intubation Conditions
MeSH Terms: interventions — Succinylcholine; Rocuronium

STUDY DESIGN:
Intervention Model Description: Randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocuronium group (Active Comparator): Rocuronium 1 mg/kg
  Interventions: Drug: Rocuronium
- Suxamethonium group (Active Comparator): Suxamethonium 1 mg/kg
  Interventions: Drug: Suxamethonium

INTERVENTIONS:
Drug: Suxamethonium — 1 mg/kg for tracheal intubation after 60 seconds
  Other Names: Succinylcholine
  Arms: Suxamethonium group
Drug: Rocuronium — 1 mg/kg for tracheal intubation after 60 seconds
  Other Names: Esmeron
  Arms: Rocuronium group

SUMMARY:
The aim of this study is to determine the proportion of excellent tracheal intubation conditions at 60 seconds after administration of either rocuronium 1.0 mg/kg or suxamethonium 1 mg/kg in patients with age ≥ 80 years during rapid sequence induction.

DETAILED DESCRIPTION:
Elderly patients are frail and susceptible to complications in the perioperative period. They are at higher risk of major morbidity and mortality and are characterized by a reduction in cardiac output, liver function and renal function. These physiological changes influence pharmacodynamics and pharmacokinetics of drugs administered during anesthesia as for example neuromuscular blocking agents (NMBA).

The number of elderly patients (>80 years) is increasing and a large proportion of these patients will require surgery and anesthesia with employment of rapid sequence induction (RSI) within the next decades. RSI and intubation is performed when there is an increased risk of pulmonary aspiration of gastric contents. Because of its fast onset time succinylcholine is often used to facilitate tracheal intubation during RSI. However, succinylcholine has certain side effects such as cardiac arrhythmia, hyperkalemia, muscle soreness, short duration of action and shorter time to desaturation.

It is therefore unknown if succinylcholine 1.0 mg/kg provides better intubating conditions compared to high dose rocuronium (1.0 mg/kg) in the elderly. In this matter, there remains a need for a study to investigate the optimal muscle relaxant during rapid sequence induction for facilitating tracheal intubation in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80
* Scheduled for surgery under general anesthesia with indication for rapid sequence induction
* American Society of Anesthesiologists physical status classification (ASA) I to IV
* Informed consent (see appendix 1)
* Body mass index (BMI) < 35 kg/m2
* Read and understand Danish

Exclusion Criteria:

* Neuromuscular disease
* Known allergy to rocuronium and/or suxamethonium
* Known hyperkalemia > 5 mM
* Previous malignant hyperthermia
* Known homozygote plasmacholinesterase gene mutation variant a or s
* Known impaired kidney function defined as estimated glomerular filtration rate (eGFR) < 30

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Intubation conditions | 60 seconds after induction of anaesthesia
  Tracheal intubating conditions according to the Fuchs-Buder scale: Excellent, good or poor depending on laryngoscopy, vocal chords and reaction to intubation,

SECONDARY OUTCOMES:
Time to tracheal intubation | within 15 minutes after administration of muscle relaxant
  • Time to tracheal intubation (from administration of muscle relaxant till correct placement of tracheal tube)
Time to TOF count 0 | within 15 minutes
  Time till no response from the nerve-stimulator after administration of muscle relaxant
First pas succes rate | within 15 minutes
  Succes of tracheal tube placement 60 seconds after administration of muscle relaxant
Intubation conditions | within 15 minutes
  Intubation conditions evaluated on the Intubation Difficulty Scale ranging from 0 (best) til 10 (worst)
Desaturation | within 15 minutes
  spO2 < 0.9
cardiac arrythmia | within 15 minutes of anesthesia
  Occurrence of new cardiac arrythmia during induction of anaesthesia (<15 minutes from administration of muscle relaxant)
sore throat | 24 hours after anaesthesia
  blinded assessment of sore throat reported by the patient on a numerical ranking scale (0 best, 10 worst)
muscle soreness | 24 hours after anaesthesia
  blinded assessment of muscle soreness reported by the patient on a numerical ranking scale (0 best, 10 worst)

CONTACTS AND LOCATIONS:
Overall Officials: Lars S Rasmussen, Study Chair — Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Department of Anaesthesiology, Pain and Respiratory Support, Rigshospitalet Glostrup, Glostrup Municipality
  - Holbæk Hospital, Holbæk

IPD SHARING:
Plan to Share IPD: No